CLINICAL TRIAL: NCT01764646
Title: Stereotactic Body Radiation Therapy for cT1c - cT3a Prostate Cancer With a Low Risk of Nodal Metastases (≤ 20%, Roach Index): a Novalis Circle Phase II Prospective Randomized Trial
Brief Title: Hypofractionated Radiation Therapy in Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Thomas Zilli (Other)
Responsible Party: Sponsor-Investigator, Thomas Zilli, Dr, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-196
Record Dates: First submitted 2012-12-20; First posted 2013-01-09 (Estimated); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Malignant Neoplasm of Prostate; Local Disease
Keywords: Prostate cancer; Radiation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Radiotherapy, Image-Guided

STUDY DESIGN:
Intervention Model Description: 5 x 7.25 Gy delivery in 2 alternative time Schedule: over 9 days every other treatment or over 28 days once a week
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 9 days (Experimental): Patients undergo extreme hypofractionated radiation therapy (Intensity modulated radiation therapy, Volumetric modulated arc therapy, Image guided radiation therapy) once a week over 28 days
  Interventions: Radiation: Intensity modulated radiation therapy; Radiation: Volumetric modulated arc therapy; Radiation: Image guided radiation therapy
- 28 days (Experimental): Patients undergo extreme hypofractionated radiation therapy (Intensity modulated radiation therapy, Volumetric modulated arc therapy, Image guided radiation therapy) other 9 days.
  Interventions: Radiation: Intensity modulated radiation therapy; Radiation: Volumetric modulated arc therapy; Radiation: Image guided radiation therapy

INTERVENTIONS:
Radiation: Intensity modulated radiation therapy — Minimize radiation doses to surrounding area
Radiation: Volumetric modulated arc therapy — Highly conformational dose distribution
Radiation: Image guided radiation therapy — Follow target by the use of fiducial markers and ERB

SUMMARY:
RATIONALE: It is not yet known whether extreme hypofractionation is equally safe and effective than standard radiation therapy in treating prostate cancer.

PURPOSE: This protocol presents a randomised phase II study aiming to investigate the tolerance and disease control of extreme hypofractionated Radiation Therapy for prostate cancer.

DETAILED DESCRIPTION:
This protocol presents a randomised phase II study aiming to investigate the tolerance and disease control of extreme hypofractionated RT for prostate cancer by delivering 5 x 7.25 Gy = 36.25 Gy over two alternative time schedules: either over 9 days (study A), or over 28 days once-a-week, the same week-day (study B).

The total dose and fractionation schedules have been chosen based on the assumption of their isoeffectivity regarding potential late rectal effects to be expected with a maximum equivalent dose of 74 Gy in 2 Gy fractions and assuming an alpha/beta = 3 Gy for the rectum.

In both arms, the prescribed dose per fraction to the urethra and the surrounding transitional zone will be dropped from 7.25 Gy to 6.5 Gy with a simultaneous integrated boost (SIB) technique. A dose of 5 x 6.5 Gy is equivalent to 31 x 2 Gy assuming an alpha/beta = 3 Gy for the urethra and equivalent to 37 x 2 Gy assuming an alpha/beta = 1.5 Gy for microscopic tumour foci in the transitional zone surrounding the urethra. The two treatment regimens chosen will each be the object of a separate phase I-II study covered by the same protocol and performed in parallel by the participating centres. Randomised assignment to either of the two studies will be introduced to avoid selection bias in treatment assignment within each centre.

OBJECTIVES:

Primary

* To determine the risk of urinary, rectal and sexual acute and late toxicities rates in patients receiving two different time schedules of extreme hypofractionated radiation therapy

  • Secondary
* To determine the Quality of life (EORTC QLQ-C30, Prostate cancer module EORTC QLQ-PR25) in patients receiving two different time schedules of extreme hypofractionated radiation therapy
* To determine the rate of local failure
* To determine in the two study arms the biochemical disease-free survival bDFS rate
* To determine in the two study arms the metastases-free survival rate
* To determine in the two study arms the disease-specific survival rate

OUTLINE:

This is a multicenter study.

Patients undergo extreme hypofractionated radiation therapy for prostate cancer by delivering 5 x 7.25 Gy = 36.25 Gy over two alternative time schedules:

Experimental Arm A: Over 9 days. Experimental Arm B: Over 28 days once-a-week, the same week-day. All patients will be followed up for at least 18 months to contribute to the analysis of the main endpoints of the study. With reference to the secondary endpoints, follow-up will be extended to 10 years.

Stopping rule: In order to avoid exposure of patients to a treatment that may be unsafe, acute GI and GU toxicity will be continuously monitored with the purpose of assisting in the decision of possibly interrupt recruitment in case of an alarming frequency.To this purpose, the procedure of Ivanova et al., 2005 will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Age: >18
* WHO performance status ≤ 2
* Any patient where prophylactic lymph node irradiation is not required, i.e. risk of nodal microscopic involvement ≤ 20% (according to Roach et al (25):

"N+ (in %) = (Gleason score - 6) x 10 + 2/3 PSA at diagnosis)"

* T-stage: cT1-cT3a.
* Previous TURP is allowed provided there is at least 8 weeks interval with radiotherapy.
* Combined hormonal treatment (Neoadjuvant-concomitant androgen deprivation, AD, for 6 months) is mandatory if two or more of the following tumour characteristics are present: ≥cT2c, Gleason 4+3, PSA >10 ng/ml, perineural invasion, and/or >1/3 of positive biopsies. RT shall be delivered between 2 and 3 months (+/- 1 week) after starting AD and according to the following chronologic sequence:

  1. Neoadjuvant AD for 2 months (30 days of bicalutamide 50mg qd, and a 3-month slow-releasing LH-RH analog to be started 15 days after initiating bicalutamide).
  2. Randomization at the end of the neoadjuvant AD period (2 months after starting AD).
  3. Planning RT (to be started within 1 month after randomization (i.e., between the 2nd and 3th month after initiating AD)
* Concomitant and adjuvant HT for 4 more months (a second 3-month slow-releasing LH-RH analog injection).

Exclusion Criteria:

* Inability to obtain a written informed consent
* Patient preference to be treated with one rather than the other treatment arm.
* WHO performance status > 2
* cT3b,cT4
* Gleason score ≥8
* Clinical N+ on metastases work-up or N+ risk >20% (Roach algorithm)
* Severe urinary obstructive symptoms (IPSS symptom index >19)
* Previous TURP less than 8 weeks before radiotherapy
* Previous prostate surgery other than TURP

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2012-09; Primary Completion 2020-12 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Tolerance to treatment | up to 5 years
  Tolerance to treatment (urinary, rectal, sexual): Acute (up to 90 days) and late (up to 5 years) toxicity follow-up according to NCI CTCAE version 3.0

SECONDARY OUTCOMES:
1. Quality of life | 9 days (Treatment arm A) or 28 days (Treatment arm B), 12 weeks, 6, 12, 18 months and yearly thereafter, up to 5 years
  Quality of life (EORTC QLQ-C30, Prostate cancer module EORTC QLQ-PR25)
2. Local failure | 9 days (Treatment arm A) or 28 days (Treatment arm B), 12 weeks, 6, 12, 18 months and yearly thereafter, up to 5 years
  Assessed by digital rectal examination (DRE). MRI or PET-CT with choline or acetate may be a confirmatory option. Biopsy confirmation is required for those patients with exclusive local failures and candidates for local salvage.
3. Biochemical disease-free survival bDFS | 9 days (Treatment arm A) or 28 days (Treatment arm B), 12 weeks, 6, 12, 18 months and yearly thereafter, up to 5 years
  Phoenix definition (PSA nadir + 2 ng/ml)
4. Metastases-free survival | 9 days (Treatment arm A) or 28 days (Treatment arm B), 12 weeks, 6, 12, 18 months and yearly thereafter, up to 5 years
  Outcomes 3 or 4 - investigations PET-CT choline
5. Disease-specific survival | 9 days (Treatment arm A) or 28 days (Treatment arm B), 12 weeks, 6, 12, 18 months and yearly thereafter, up to 5 years
  Alive/dead status, date and cause of death and prostate cancer disease status (outcomes 3/4 and 5).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zilli, Dr, Principal Investigator — University Hospital, Geneva
Locations (9):
- Onze Lieve Vrouwziekenhuis, Aalst, Belgium
- University Hospital, Turku, Finland
- Sheba Medical Center, Ramat Gan, Israel
- VU University Medical Center, Amsterdam, Netherlands
- Portuguese Institut of Oncology, Porto, Portugal
- Spain (2):
  - Teknon Oncologic Institute, Barcelona
  - Hospital Universitario Sanchinarro, Madrid
- University Hospital, Geneva, Switzerland
- Neolife Medical Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
No plan to share participant data for now